CLINICAL TRIAL: NCT05924672
Title: Efficacy of Ra-223 in PSMA PET Optimally Selected Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23923; NCI-2023-04656 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223; radium Ra 223 dichloride; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Glutamate Carboxypeptidase II; Technetium Tc 99m Medronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (NaF PET/CT/MDP, Ra-223, PSMA PET) (Experimental): Patients undergo NaF PET/CT or MDP scan within 45 days prior to cycle 1 day 1. Patients then receive standard of care Ra-223 IV on day 1 of each cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo PSMA PET/CT over 45-60 minutes between 30-60 days after the last dose of Ra-223. Patients also undergo collection of blood samples during screening, on day 1 of every Ra-223 cycle, and at 30 days after the last dose of Ra-223. Patients may also undergo NaF PET/CT or MDP scans during Ra-223 treatment as clinically indicated, and/or CT scans during screening and Ra-223 treatment as clinically indicated.
  Interventions: Drug: Radium-223; Procedure: PSMA Positron Emission Tomography (PET) Scan; Drug: Technetium Tc 99M Medronate

INTERVENTIONS:
Drug: Radium-223 — Given IV
  Other Names: Ra-223; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; Xofigo
Procedure: PSMA Positron Emission Tomography (PET) Scan — Undergo PSMA PET/CT
  Other Names: Prostate-specific Membrane Antigen (PSMA) PET; PSMA PET
Drug: Technetium Tc 99M Medronate — Undergo MDP
  Other Names: (99m)Tc-Medronate, 121524-79-6; 99mTc-MDP; TechneScan MDP; Technetium Tc 99m Methylene Diphosphonate

SUMMARY:
This phase II trial studies how well prostate-specific membrane antigen (PSMA) positron emission tomography (PET) scans (in combination with bone scans) work in selecting patients for Ra-223 radiation therapy that have castration-resistant prostate cancer that has spread from where it first started (primary site) to the bones (bone metastasis). Ra-223 is a type of therapy that emits radiation. Radiation gives off energy which can kill tumor cells and other cells that may support the tumor cells. Ra-223 is given by infusion into the veins, where it is absorbed by the bones. PSMA PET is a type of scan used to detect prostate cancer tumors. PSMA is a radioactive tracer that binds to a specific protein that is found on prostate tumor cells. The PSMA tracer shows the areas on the PET scan where tumor cells are active. A PET scan uses a special camera to detect the energy given off from radioactive tracers (such as PSMA) to make detailed pictures of areas where the tracer accumulates in the body. The PET scan is often combined with a magnetic resonance imaging (MRI) or computed tomography (CT) scan, which helps to map the locations where PSMA has accumulated. PSMA PET scans may be able to select patients that will benefit the most from Ra-223 treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the PSA50 response rate of participants treated with radium Ra 223 dichloride (Ra-223).

SECONDARY OBJECTIVES:

I. To determine the median overall survival (mOS) of participants treated with Ra-223.

II. To determine the PSA30 response rate of participants treated with Ra-223. III. To determine the time to the first skeletal symptomatic event. IV. To characterize the safety profile of Ra-223 treatment. V. To compare the lesion based PSMA PET response based on sodium fluoride (NaF) PET/technetium Tc-99m medronate (MDP) single photon emission computed tomography (SPECT) uptake.

EXPLORATORY OBJECTIVES; I. To compare the PSA response stratified by PSMA PET tumor volume. II. To determine the location of progression by location. III. Safety on subsequent treatment with PSMA radioligand therapy (RLT).

OUTLINE:

Participants undergo NaF PET/CT or MDP scan within 45 days prior to standard of care (SOC) Ra-223 intravenously (IV). Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Participants then undergo a PSMA PET/CT between 30-60 days after the last dose of Ra-223. Participants also undergo collection of blood samples during screening, on the first day of every Ra-223 cycle, and at 30 days after the last dose. Participants may also undergo a NaF PET/CT or MDP scan during treatment as clinically indicated, and/or CT scans during screening and treatment as clinically indicated.

After completion of Ra-223 treatment, participants are followed up at 30 days, and then every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male participants >= 18 years of age on the day of signing informed consent
* Castrate level of serum testosterone at study entry (< 50 ng/dL), checked within three months of enrollment
* Patient is a candidate for standard of care Ra-223 therapy
* Bone only disease on PSMA PET using a Food and Drug Administration (FDA) approved PSMA targeted PET radiopharmaceutical

  * Note: Nodal disease on PSMA PET that is less than 1 cm in short axis and without evidence of change in size over the past six months on conventional imaging is allowed
  * Positivity on PSMA PET is defined as uptake greater than the liver that is not attributable to physiologic activity
* Histologically confirmed prostate adenocarcinoma that is progressive by Prostate Cancer Working Group 3 (PCWG3) criteria at the time of study entry
* Prior progression on at least one second generation androgen signaling inhibitor including abiraterone, apalutamide, darolutamide, and/or enzalutamide
* Platelets > 100,000/microliter (mcL)
* Hemoglobin (Hgb) > 9.0 g/dL
* White blood cells (WBC) > 2.5
* Albumin > 3.0 g/dL
* Adverse events related to prior anti-cancer treatment must have recovered to =< Grade 2
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* For patients who have partners of childbearing potential: Partner and/or patient must use a method of birth control with adequate barrier protection, deemed acceptable by the principal investigator during the study and for 3 months after last study drug administration
* Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior treatment with Lutetium-177 (177Lu)-PSMA-617, Radium-223, Strontium-89, Samarium-153, Rhenium-186, Rhenium-188
* Prior exposure to taxane-based chemotherapy.

  * Note: Exposure is defined as two or more cycles of taxane-based agents
* Any systemic anti-cancer therapy (e.g., chemotherapy, immunotherapy or biological therapy, including monoclonal antibodies) within 21 days prior to the first day of treatment
* Greater than 75% bone involvement, based on PSMA PET
* Presence of visceral metastases, untreated central nervous system metastases, or untreated epidural or spinal cord involvement
* Prior treatment with radioligand therapy
* Blood transfusion within past 45 days
* Any condition that, in the opinion of the Principal Investigator, would impair the patient's ability to comply with study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
PSA50 response rate | Up to 6 months
  The proportion of patients who achieve a greater than 50% decline from baseline prostate specific antigen (PSA) (PSA50) drawn prior to C1D1, at any point in the treatment course, will be descriptively reported along with 95% binomial confidence interval. It will be compared with the historical control by binomial test. A confirmation repeat PSA will be drawn after the initial PSA50 response to confirm the result. A PSA50 will only be counted if two PSA showing a 50% decline are measured.

SECONDARY OUTCOMES:
PSA30 response rate | Up to 6 months
  The proportion of patients who achieve a greater than 30% decline from baseline PSA (PSA30) drawn prior to cycle 1 day 1 (C1D1), at any point in the treatment course, will be descriptively reported along with 95% binomial confidence interval. It will be compared with the historical control by binomial test.
Overall Survival | Up to 2 years
  Overall survival The time to event will be defined by the duration from the first date of study therapy to date of death from any cause. We will estimate the survival function using the Kaplan-Meier method, and obtain its 95% confidence bands over the survival times. The median overall survival time and 95% confidence interval of it will be derived from the estimated survival functions.
Time to first skeletal symptomatic event | Up to 30 days after the last dose of Ra-223 treatment
  The time to the first skeletal symptomatic event will measure the time to the first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, or requirement for radiation therapy to relieve bone pain, whichever occurs first. We will also estimate the survival function using the Kaplan-Meier method, and obtain its 95% confidence bands over the survival times. The median survival time and 95% confidence interval of it will be derived from the estimated survival functions.
Proportion of participants reporting treatment-related adverse events | Up to 30 days after the last dose of Ra-223 treatment
  The incidence and severity of adverse events related to study treatment will be descriptively reported using CTCAE v5.0.
Compare the lesion based PSMA PET response based on paired NaF PET / MDP uptake | Up to 30 days after the last dose of Ra-223 treatment
  Up to five lesions per patient will be measured by a board certified nuclear medicine physician. For each lesion the maximum SUV (SUVmax) will be measured on PSMA PET and NaF PET. Additionally, the SUVmax on the end of study PSMA PET will also be measured. As there is an underestimation of uptake on MDP bone scan compared to PET, we will multiply the uptake measured on MDP SPECT by 2.3 to correct for the differences in recovery coefficients between the two imaging technologies based on prior comparisons. The percent change in the PSMA PET uptake between baseline and end of study will be measured. A Spearman's rank correlation will be used to compare the baseline NaF uptake for each lesion with the percent change of PSMA PET SUVmax.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No